CLINICAL TRIAL: NCT03517800
Title: Surgical Management of Intractable Postpartum Haemorrhage When Arterial Embolization Can't be Performed : Feasibility an Complications.
Brief Title: Surgical Management of Postpartum Haemorrhage Without Embolization
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0259
Record Dates: First submitted 2017-10-12; First posted 2018-05-07 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2017-10

CONDITIONS: Postpartum Hemorrhage; Second Line Management; Uterine Arteries Embolization; Surgical Management of Haemorrhage
Keywords: Embolization; surgery; hysterectomy; arterial ligation
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Arterial embolization and/or surgical management. — Arterial embolization and/or surgical management.

SUMMARY:
Postpartum haemorrhage is the main cause of maternal mortality. The aim of investigators' study was to evaluate the practice of hemostatic surgery (arterial ligation, uterine compression or hysterectomy) when the embolization of uterine arteries wasn't be performed.

ELIGIBILITY:
Inclusion criteria:

* Age over 18
* Postpartum haemorrhage
* Necessity of second line management
* No embolization performed
* Necessity of surgical management after embolization

Exclusion criteria:

* Unnecessity of second line management
* Management by only embolization
* Incomplete medical files

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with postpartum haemorrhage with a surgical management in a type III universitary maternity.
Sampling Method: Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Frequency of each type of surgical management | at delivery
  Frequency of each type of surgical management

SECONDARY OUTCOMES:
Number of surgical interventions | at delivery
  Number of surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOULOT, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC